CLINICAL TRIAL: NCT04667897
Title: A Randomized, Double Masked, Multicenter, Phase II Study Assessing the Safety and Efficacy of 601 Versus Ranibizumab in Patients With Visual Impairment Due to Macular Edema Secondary to Branch Retinal Vein Occlusion (BRVO)
Brief Title: 601 Versus Ranibizumab in Patients With Branch Retinal Vein Occlusion (BRVO)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SSGJ-601-BRVO-II-01
Record Dates: First submitted 2020-12-08; First posted 2020-12-16 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2022-07

CONDITIONS: Branch Retinal Vein Occlusion
Keywords: VEGF; BRVO; antibody
MeSH Terms: conditions — Retinal Vein Occlusion | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 601 1.25mg (Experimental)
  Interventions: Drug: 601 1.25mg
- Ranibizuman 0.5 mg (Experimental)
  Interventions: Drug: Ranibizuman 0.5 mg

INTERVENTIONS:
Drug: 601 1.25mg — Solution for injection (intravitreal use)
  Other Names: Drug 601
  Arms: 601 1.25mg
Drug: Ranibizuman 0.5 mg — Solution for injection (intravitreal use)
  Other Names: Lucentis
  Arms: Ranibizuman 0.5 mg

SUMMARY:
To evaluate the safety and efficacy of intravitreal recombinant humanized anti-VEGF monoclonal antibody in patients with visual impairment due to macular edema secondary to BRVO

DETAILED DESCRIPTION:
Following a 14-day maximum screening period, patients will be randomized and followed for approximately 52 weeks. Treatment visits will be scheduled in 4-week intervals. After 6 initial monthly injections of 601 or ranibizumab (loading phase), subjects will enter an individualized flexible treatment (IFT) phase (week 24 to week 48). During the IFT phase, an assessment of disease stability will be performed at each monthly visit and subjects will receive either an injection or not. Safety and efficacy outcomes will continue to be evaluated up to a period of 52 weeks unless the patient is withdrawn or discontinues the study.

ELIGIBILITY:
Inclusion Criteria:

* Sign informed consent form and willing to be visited at the time specified in the trial
* Male or Female, at least 18 years of age
* The study eye must meet the following criteria

  1. Diagnosed with macular edema secondary to Branch retinal vein occlusion (BRVO) or Hemiretinal vein occlusion (HRVO) within 12 months
  2. BCVA score between 78 and 19 letters, inclusive, using ETDRS visual acuity testing charts (approximate Snellen equivalent of 20/32 to 20/400)
  3. CRT ≥ 250μm
  4. No optometric media opacity and pupil abnormal
* BCVA score ≥ 34 letters in the fellow eye, using ETDRS visual acuity testing charts (approximate Snellen equivalent of 20/200)

Exclusion Criteria:

For Study Eye:

* Concomitant conditions or ocular disorders in the study eye at screening or baseline which could, in the opinion of the investigator, prevent response to study treatment or may confound interpretation of study results, compromise visual acuity or require medical or surgical intervention during the first 12-month study period (e.g. scarring, fibrosis or atrophy of the fovea, dense subfoveal hard exudates, significant hemorrhage obscuring the macular, vitreous hemorrhage, vitreomacular traction, retinal vascular occlusion other than BRVO or HRVO, retinal detachment, macular hole, or age-related macular degeneration，choroidal neovascularization of any cause, diabetic retinopathy (except mild non-proliferative) and diabetic macular edema)
* iris, chamber angle neovascularization or retinal, optic disc neovascularization
* Previous use of intraocular or periocular steroids within 3 months prior to baseline, or previous use of dexamethasone intravitreal implant within 6 months prior to baseline
* Macular laser photocoagulation (focal/grid)，panretinal laser photocoagulation，vitrectomy，radial optic neurotomy arteriovenous sheathotomy，trabeculectomy or keratoplasty in the study eye at any time prior to baseline. Local laser photocoagulation, YAG laser treatment or any other ocular surgeries (e.g. cataract surgery ) in the study eye within 3 months prior to the baseline
* During the screening period, the BCVA is >10 letters improved (the BCVA detected within 24 hours before the administration at day 0 compared with the BCVA at the screening)
* Aphakia (except IOL) or posterior capsular defect (except YAG posterior capsulotomy after intraocular lens implantation surgery)

For Any Eye:

* Any eye has active ocular infections (e.g. blepharitis, conjunctivitis, keratitis, scleritis, uveitis, endophthalmitis)
* Uncontrollable glaucoma (defined as intraocular pressure after antiglaucoma therapy>= 25 mm Hg), or the cup/disk ratio >0.8 in the study eye
* History of intravitreal use of anti-VEGF drugs (e.g. ranibizumab，bevacizumab，aflibercept, conbercept, etc.) in any eye within 3 months prior to baseline

General Exclusion Criteria:

* History of allergy to fluorescein sodium and allergies to protein products for treatment or diagnosis
* History of stroke (cerebrovascular accident), myocardial infarction, active disseminated intravascular coagulation or pronounced bleeding tendency in the past 6 months prior to baseline
* Diagnosed systemic immune diseases (e.g. ankylosing spondylitis, systemic lupus erythematosus, Behcet's disease, rheumatoid arthritis, scleroderma etc.)
* any uncontrolled clinical problem (e.g. AIDS, active hepatitis, serious mental, neurological, cardiovascular, respiratory and other systemic diseases or malignant tumors, etc.). Malignant tumors with no metastasis or recurrence within 5 years or cancers in situ cancers are not excluded.
* Uncontrolled blood pressure control (defined as systolic blood pressure > 160 mmHg or diastolic pressure > 100 mmHg after antihypertensive medication
* History of surgery (except for healed minimally invasive surgery) and/or currently have unhealed wounds, moderate to severe ulcers, fractures, etc. within 1 month prior to baseline
* History of system use of anti-VEGF drugs (e.g. bevacizumab) within 3 months prior to baseline

Laboratory Exclusion Criteria:

* Liver dysfunction (ALT or AST is 2 times higher than the upper limit of normal value in the local laboratory). Renal function impairment (Cr is 1.5 times higher than the upper limit of normal values in the local laboratory)
* Abnormal coagulation function (prothrombin time >= the upper limit of normal value for 3 seconds) and activated partial thromboplastin time >= the upper limit of normal value for 10 seconds);

Other Exclusion Criteria:

* Non-use of effective contraception during childbearing age (except for women with spontaneous admonishment of more than 12 months)
* Pregnancy and lactation women
* Participation in clinical trials of any drug (except vitamins and minerals) or medical devices in the past 1 month or 5 half-lifes if the drug has a long half-life >1 month prior to baseline;
* Researchers think it needs to be ruled out

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-01-28 (Actual); Primary Completion 2022-07-13 (Actual); Study Completion 2022-07-13 (Actual)

PRIMARY OUTCOMES:
Change from baseline in best-corrected visual acuity (BCVA) at Week 24 | Baseline to Week 24
  Assessed with ETDRS visual acuity testing charts.

SECONDARY OUTCOMES:
Change from baseline in BCVA by visit up to Week 12 and Week 52 | Baseline, Week 12 and Week 52
  Assessed with ETDRS visual acuity testing charts.
Proportion of study eyes with a gain ≥ 5, 10 and 15 letters in BCVA by at Week 12, Week 24 and Week 52 compared to baseline | Baseline, Week 12, Week 24 and Week 52
  Assessed with ETDRS visual acuity testing charts.
Average Change of BCVA From Baseline to Week 4 Through Week 52 | Baseline to Week 52
  Assessed with ETDRS visual acuity testing charts.
Average Change of BCVA From Baseline to Week 28 Through Week 52 | Week 28 to Week 52
  Assessed with ETDRS visual acuity testing charts.
Change from baseline in central retina thickness (CRT) at Week 12, Week 24 and Week 52 | baseline, Week 12, Week 24 and Week 52
  OCT (optical coherence tomography) was used to assess central retina thickness (CRT) representing the average retinal thickness of the central 1 mm diameter subfield around the foveal center.
Number of injections from baseline to Week 52 | baseline to Week 52
  Number of administered injections
Number of injections between Week 24 to Week 52 | Week 24 to Week 52
  Number of administered injections
Incidence of ocular and non-ocular AEs up to Week 52 | Baseline to Week 52
  Incidence of ocular and non-ocular AEs
Blood concentrations of 601 at Baseline, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24，Week 36 and Week 52 | Baseline, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24，Week 36 and Week 52
  Steady-state blood concentrations of 601
Blood concentrations of VEGF at Baseline, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24，Week 36 and Week 52 | Baseline, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24，Week 36 and Week 52
  Detection of VEGF blood concentration.
Immunogenicity of 601 at Baseline, Week 4, Week 12, Week 24, Week 36 and Week 52 | Baseline, Week 4, Week 12, Week 24, Week 36 and Week 52
  Detection of blood Anti-drug antibody (ADA) status. If ADA was positive, Neutralization antibody (Nab) will be tested.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Dai, Bachelor, Principal Investigator — Beijing Hospital
Locations (1):
- BeiJing Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No